CLINICAL TRIAL: NCT00812591
Title: Evaluation of a Novel Method for Integrating Insulin Delivery and Glucose Sensing in Subcutaneous Tissue for the Treatment of Type-1 Diabetic Patients
Brief Title: Integrating Insulin Delivery and Glucose Sensing in Subcutaneous Tissue for the Treatment of Type-1 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Stefan Korsatko, MD, MD, Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ZIG26
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucose Tolerance Test; Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: OGTT and CLAMP — Oral Glucose Tolerance Test (OGTT):
  Oral glucose tolerance test combined with subcutaneous insulin delivery and glucose sampling using a single microdialysis or microperfusion probe.
  Hyperinsulinemic euglycemic clamp (CLAMP):
  Hyperinsulinemic euglycemic clamp with simultaneous subcutaneous insulin delivery and glucose sampling using microdialysis and microperfusion probe.

SUMMARY:
The study seeks to use microdialysis and microperfusion techniques to assess the feasibility of combining insulin delivery and glucose sensing at a single subcutaneous tissue site.

DETAILED DESCRIPTION:
Current treatment of in type 1 diabetes comprises the measurement of glucose in capillary blood obtained by fingersticking and administration of exogenous insulin in the form of a subcutaneous bolus injection or subcutaneous infusion. This treatment could be simplified if there were a stable ratio between blood glucose concentration and tissue glucose level at the site of insulin delivery so that tissue glucose levels could be used to estimate blood glucose levels, thereby circumventing the need for fingerstick blood glucose monitoring.

The aim of this study is to ascertain whether a stable ratio between the blood glucose concentration and the glucose levels at the tissue site of insulin infusion exists when this tissue site is exposed to variable insulin infusion rates. To achieve this, microdialysis and microperfusion probes are applied in healthy and type 1 diabetic subjects to perform insulin delivery and glucose sampling at the same adipose tissue site during euglycemic clamps and oral glucose tolerance tests.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus patients aged 18 - 65
* Healthy subjects aged 18 - 65
* Informed consent obtained before any trial-related activities.

Diabetic subjects:

* C-peptide negative (≤ 0.05 nmol/L)
* HbA1c (glycosylated haemoglobin A1c) < 10%

Exclusion Criteria:

* Severe diabetic complications (e.g., proliferative retinopathy, severe nephropathy)
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods
* Subject with mental incapacity or language barriers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Ratio between the plasma glucose level and the glucose concentration at the subcutaneous insulin delivery site | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz, Internal Medicine, Endocrinology and Nuclear Medicine
Locations (1):
- Medical University of Graz, Graz, Styria, Austria